CLINICAL TRIAL: NCT02834507
Title: A Double-blind, Randomised, Placebo- and Active-controlled, Cross-over Study to Investigate the Effect of Two Multiple-dose Regimens of BIA 3-202 on the Pharmacokinetics and Motor Response of Levodopa, and on the Erythrocyte Comt Activity in Parkinson's Disease Patients
Brief Title: Effect of Two Multiple-dose Regimens of BIA 3-202 on the Pharmacokinetics and Motor Response of Levodopa, and on the Erythrocyte Comt Activity in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-3202-201
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson's Disease (PD)
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone; entacapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): In each treatment period, patients received, in a double-blind manner, 1 capsule of investigational product (nebicapone 75 mg, nebicapone 150 mg, entacapone 200 mg or placebo, according to the treatment sequence), concomitantly with each levodopa/carbidopa (Sinemet®) dose patient used to take.
  Interventions: Drug: Placebo; Drug: Sinemet®
- Nebicapone 75 mg (Experimental): In each treatment period, patients received, in a double-blind manner, 1 capsule of investigational product (nebicapone 75 mg, nebicapone 150 mg, entacapone 200 mg or placebo, according to the treatment sequence), concomitantly with each levodopa/carbidopa (Sinemet®) dose patient used to take.
  Interventions: Drug: BIA 3-202; Drug: Sinemet®
- Nebicapone 150 mg (Experimental): In each treatment period, patients received, in a double-blind manner, 1 capsule of investigational product (nebicapone 75 mg, nebicapone 150 mg, entacapone 200 mg or placebo, according to the treatment sequence), concomitantly with each levodopa/carbidopa (Sinemet®) dose patient used to take.
  Interventions: Drug: BIA 3-202; Drug: Sinemet®
- Entacapone 200 mg (Active Comparator): In each treatment period, patients received, in a double-blind manner, 1 capsule of investigational product (nebicapone 75 mg, nebicapone 150 mg, entacapone 200 mg or placebo, according to the treatment sequence), concomitantly with each levodopa/carbidopa (Sinemet®) dose patient used to take.
  Interventions: Drug: Comtan®; Drug: Sinemet®

INTERVENTIONS:
Drug: Placebo — Matching placebo capsules
  Arms: Placebo
Drug: BIA 3-202 — Capsules containing nebicapone 75 mg or 150 mg
  Other Names: Nebicapone
  Arms: Nebicapone 150 mg; Nebicapone 75 mg
Drug: Comtan® — Capsules containing entacapone 200 mg
  Other Names: Entacapone
  Arms: Entacapone 200 mg
Drug: Sinemet® — levodopa/carbidopa (Sinemet®) dose patient used to take
  Other Names: levodopa/carbidopa

SUMMARY:
The purpose of this study is to determine the effect of two different multiple-dose regimens of nebicapone in comparison to placebo and entacapone 200 mg on the pharmacokinetics of levodopa in Parkinson's Disease (PD) patients.

DETAILED DESCRIPTION:
STUDY DESIGN AND METHODOLOGY:

This was a multicentre, randomised, double-blind, placebo- and active-controlled, four-way crossover study. The study consisted of 4 treatment periods in at least 16 patients with PD treated with standard release levodopa/carbidopa (Sinemet®). Patients were randomly assigned to treatment with placebo, nebicapone 75 mg, nebicapone 150 mg or entacapone 200 mg (Comtan®) in 4 different sequences.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed before screening activities.
2. Male or female aged between 30 and 75 years, inclusive.
3. A diagnosis of PD according to the UK PDS Brain Bank diagnostic criteria (bradykinesia and at least one of the following: muscular rigidity, rest tremor and postural instability).
4. Predictable signs of end-of-dose "wearing-OFF" phenomenon (end-of-dose deterioration) despite "optimal" levodopa/carbidopa therapy.
5. At least 60 minutes of daily OFF time in the two days prior to the randomisation visit day.
6. Been treated with levodopa/carbidopa for at least 1 year prior to randomisation with clear clinical improvement.
7. Been treated with a stable regimen of 3 to 6 daily doses of standard release levodopa/carbidopa (4:1 ratio) per day within at least 4 weeks prior to randomisation, although a bedtime dose of slow-release formulation is permitted.
8. Concomitant anti-Parkinsonian medication (other than apomorphine and entacapone) in stable doses for at least 4 weeks prior to randomisation.
9. Able to keep reliable ON/OFF charts (diaries), alone or with caregiver assistance.
10. Laboratory results acceptable by the investigator (not clinically significant for the well-being of the patient or for the purpose of the study).
11. Women: Post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation. In case of woman of childbearing potential, patient had to present a serum B-hCG test consistent with a non-gravid state and had to agree to remain abstinent or use effective contraceptive methods.

Exclusion Criteria:

1. Non-idiopathic parkinsonism (atypical parkinsonism, symptomatic parkinsonism, Parkinson-plus syndrome).
2. Treated with levodopa/benserazide, or with levodopa/carbidopa in a 10:1 ratio, or with levodopa/carbidopa in a controlled-release form during day-time.
3. Major depressive episode within 6 months prior to randomisation.
4. Treated with entacapone, neuroleptics, monoamine oxidase inhibitors (except selegiline not exceeding 10 mg/day) or antiemetics (except domperidone) within one month prior to randomisation.
5. Treated with apomorphine within 7 days prior to randomisation.
6. Treated with any investigational product within 2 months prior to randomisation (or within 5 half-lives, whichever is longer).
7. A psychiatric or any medical condition that might place him/her at increased risk or interfere with assessments.
8. Previous use of nebicapone or participation in a clinical study with nebicapone.
9. Known hypersensitivity to any of the ingredients of the investigational products.
10. A history of abuse of alcohol, drugs or medications within the last 2 years.
11. A clinically relevant ECG abnormality. Patient could only be randomised if the ECG was normal or, if abnormal, the abnormality was mild and not considered to be clinically relevant.
12. A history or current evidence of heart disease, including but not limited to myocardial infarction, angina, congestive heart failure and cardiac arrhythmia.
13. Unstable concomitant disease being treated with changing doses of medication.
14. A history or current evidence of any relevant disease in the context of this study, i.e., with respect to the safety of the subject (e.g., hepatic impairment) or related to the study conditions.
15. A test positive for the human immunodeficiency viruses (HIV) 1 or 2 antibodies, hepatitis B surface antigen (HBs Ag) or hepatitis C antibody (HCV Ab).
16. Donated or received blood or blood products within 3 months prior to randomisation.
17. Pregnant or breast feeding.
18. Any other condition or circumstance that, in the opinion of the investigator, may compromise the patient's ability to comply with the study protocol.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentrations (Cmax) | pre-dose, 30 min, 60 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h and 24 h post dose
  Levodopa pharmacokinetic parameters following administration of nebicapone 75 mg (n=16), nebicapone 150 mg (n=18), entacapone 200 mg (n=18) or placebo (n=17) concomitantly with Sinemet®
time to Cmax (tmax) | pre-dose, 30 min, 60 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h and 24 h post dose
  Levodopa pharmacokinetic parameters following administration of nebicapone 75 mg (n=16), nebicapone 150 mg (n=18), entacapone 200 mg (n=18) or placebo (n=17) concomitantly with Sinemet®
Area under the plasma concentration-time curve from dosing until 6 h after (AUC0-6) | pre-dose, 30 min, 60 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h and 24 h post dose
  Levodopa pharmacokinetic parameters following administration of nebicapone 75 mg (n=16), nebicapone 150 mg (n=18), entacapone 200 mg (n=18) or placebo (n=17) concomitantly with Sinemet®
Apparent elimination half-life (t1/2) | pre-dose, 30 min, 60 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h and 24 h post dose
  Levodopa pharmacokinetic parameters following administration of nebicapone 75 mg (n=16), nebicapone 150 mg (n=18), entacapone 200 mg (n=18) or placebo (n=17) concomitantly with Sinemet®

IPD SHARING:
Plan to Share IPD: Undecided